CLINICAL TRIAL: NCT01220648
Title: An Open Label, Nonrandomized, Single-center, Phase I Trial of Pretreated Philadelphia Chromosome Positive (Ph+) Chronic Myeloid Leukemia Patients in Chronic Phase (CML-CP) With Nilotinib in Combination With Low Dose Interferon-alpha (IFN) - NICOLI Study -
Brief Title: Determining the Maximum Tolerated Dose of Low Dose Interferon-alpha in Conjunction With Nilotinib in Pretreated Philadelphia Chromosome Positive (Ph+) Chronic Myeloid Leukemia Patients in Chronic Phase (CML-CP)
Acronym: NICOLI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ADE10; 2010-022006-40 (EudraCT Number)
Record Dates: First submitted 2010-10-06; First posted 2010-10-14 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; interferon alfa; nilotinib; combination; CML; Philadelphia chromosome positive (Ph+) chronic myeloid leukemia patients in chronic phase (CML-CP) after switch from previous CML treatment
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Interferon-alpha

ARMS (1):
- Nilotinib in conjunction with low dose interferon alfa (Experimental)
  Interventions: Drug: Nilotinib, interferon-alfa

INTERVENTIONS:
Drug: Nilotinib, interferon-alfa
  Other Names: AMN107

SUMMARY:
This study will assess the maximum tolerated dose of low dose interferon in conjunction with nilotinib in pretreated Philadelphia chromosome positive (Ph+) chronic myeloid leukemia patients in chronic phase (CML-CP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic myeloid leukemia in chronic phase (CML-CP) at screening
* Initial diagnosis of CML cytogenetically confirmed by the presence of the Ph+ metaphases from the bone marrow
* Patients who have been treated with nilotinib for a minimum of 6 months (1 month represents 28 days) after switch from previous CML treatments
* Patients who have been treated with stable dosing of 2x400mg nilotinib within the last month before start of study treatment
* No grade 3-4 CTC toxicities on nilotinib alone in the last month preceding the start of the study regimen

Exclusion Criteria:

* Patients who are considered Ph- because they do not have a confirmed cytogenetic diagnosis of the t(9;22) translocation in their bone marrow metaphases
* Evidence of a point mutation within the BCR-ABL gene leading to a clinically relevant amino acid exchange in the kinase domain at position T315 (gatekeeper mutation T315I)
* Impaired cardiac function
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of Clinically significant adverse events or abnormal laboratory values (dose-limiting toxicities) unrelated to disease progression, intercurrent illness, or concomitant medications on the combination treatment | 12 months

SECONDARY OUTCOMES:
Rate of major cytogenetic response (MCyR) at 6 and 12 months | 12 months
Rate of complete cytogenetic response (CCyR) at 6 and 12 months | 12 months
Rate of major molecular response (MMR) at 12 months | 12 months
Safety profile of nilotinib in combination with interferon alfa, i.e. the number of dose limiting toxicities (DLT) for each interferon alfa dose level | 12 months
Progression-free survival (PFS) | 12 months
Event-free survival | 12 months
Overall survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Leipzig, Germany

REFERENCES:
- [Background] Guilhot F, Roy L, Saulnier PJ, Guilhot J. Interferon in chronic myeloid leukaemia: past and future. Best Pract Res Clin Haematol. 2009 Sep;22(3):315-29. doi: 10.1016/j.beha.2009.10.005. PMID 19959083